CLINICAL TRIAL: NCT06920329
Title: An Exploratory Clinical Study Evaluating the Impact of Interferon Consolidation Therapy on Intrahepatic cccDNA Levels in Chronic Hepatitis B Patients Who Achieved Clinical Cure With Peginterferon α-2b Therapy.
Brief Title: Effects of Peginterferon Consolidation Therapy on Hepatic cccDNA Dynamics in CHB Patients Achieving Clinical Cure.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liang Huiqing, Chief physician, Xiamen Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024K04701
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Chronic Hepatitis b
Keywords: Peginterferon α-2b injection; cccDNA; pgRNA
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peginterferon α-2b based group (Experimental)
  Interventions: Drug: Peginterferon α-2b based injection

INTERVENTIONS:
Drug: Peginterferon α-2b based injection — Peginterferon α-2b injection, 180 μg administered subcutaneously in the abdomen or thigh once weekly, with regular follow-up for HBV recurrence. Patients will be followed up every 12 weeks.

SUMMARY:
This is a single-center, prospective, exploratory clinical study. The study plans to enroll 30 chronic hepatitis B (CHB) patients which achieved HBsAg clearance based peginterferon α-2b treatment. Eligible subjects will receive either 12-24 weeks interferon consolidation therapy (180μg administered subcutaneously in the abdomen or thigh once weekly) or not according to physician's recommendation and patient's preference, with regular follow-up for HBV recurrence. Patients will be followed up every 12 weeks. The study will evaluate changes in intrahepatic covalently closed circular DNA (cccDNA) and peripheral blood HBV pregenomic RNA (pgRNA) levels after achieving HBsAg clearance.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily enroll in the study, able to understand and voluntarily sign the informed consent form;
* Aged 18-65 years (inclusive), no gender restriction;
* A history of HBsAg positivity for at least 6 months or other evidence suggesting chronic hepatitis B;
* First observed clinical cure after treatment with peginterferon α-2b (PegIntron®), either as monotherapy or in combination with NAs, defined as serum HBsAg negative (<0.05IU/ml), HBV DNA undetectable (HBV DNA<20IU/ml), and HBeAg negative, within a 4-week window from the first observed day of clinical cure at the time of screening;
* Agreement to undergo two liver biopsies during the study;
* Negative pregnancy test within 24 hours before the first liver biopsy (for childbearing-age females); and subjects (both male and female) should use effective contraception during the study period.

Exclusion Criteria:

* Lactating women;
* Evidence of acute severe liver injury: such as ALT > 10 ULN, or significantly elevated ALT with significantly elevated bilirubin;
* Evidence of decompensated liver disease: such as ascites, esophageal varices rupture bleeding, sepsis, hepatic encephalopathy, hepatorenal syndrome, etc.; or history of decompensated cirrhosis;
* Evidence of hepatocellular carcinoma;
* Prothrombin time (PT) or INR > ULN;
* Participation in other interventional trial studies within 3 months before screening or other conditions deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in intrahepatic cccDNA and peripheral blood pgRNA levels | baseline to week48
Clearance rate of intrahepatic cccDNA | week48

SECONDARY OUTCOMES:
Correlation between changes in intrahepatic cccDNA levels and interferon consolidation therapy | baseline to week48
Correlation between changes in peripheral blood pgRNA levels and interferon consolidation therapy | baseline to week48
Correlation between intrahepatic cccDNA clearance and interferon consolidation therapy | week48
Changes in intrahepatic cccDNA levels | baseline to week48
Changes in intrahepatic HBsAg levels | baseline to week48
intrahepatic HBsAg clearance rate | baseline、week48
Histopathological scores in hepatic inflammation and fibrosis | baseline、week48
Recurrence rate | baseline to week48
Adverse Event#AE# | baseline to week48

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Liang, Ph.D, Principal Investigator — Xiamen Hospital of Traditional Chinese Medicine
Locations (1):
- Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian, China